CLINICAL TRIAL: NCT02378389
Title: A Phase I Study of Pyrotinib In Combination With Docetaxel In Patients With HER2 Positive Advanced Gastric Cancer
Brief Title: Study Evaluating Pyrotinib/Pyrotinib in Combination With Docetaxel in Patients With HER2+ Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLTN-Id
Record Dates: First submitted 2015-02-11; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: HER2 Positive Gastric Cancer
MeSH Terms: interventions — pyrotinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pyrotinib/Pyrotinib with Docetaxel (Experimental): Subjects would be treated with Pyrotinib (Part 1) or Pyrotinib with Docetaxel (Part 2). A subject is only allowed to participant in one part of this trial.
  Interventions: Drug: Pyrotinib/Pyrotinib with Docetaxel

INTERVENTIONS:
Drug: Pyrotinib/Pyrotinib with Docetaxel — Pyrotinib oral daily, 240 mg, 320 mg, 400 mg.... Docetaxel i.v. once every 21 days.

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both EGFR and HER-2 receptors. This study is designed to evaluate the safety and tolerability of Pyrotinib or Pyrotinib in combination with Docetaxel in patients with HER2 positive advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤70 years.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* At least one measurable lesion exists.(RECIST 1.1).
* Histologically or cytologic confirmed HER2 positive advanced gastric cancer (including adenocarcinoma of esophageal-gastric junction), with clinical phase III/IV.
* No severe impairment of liver and kidney function, required laboratory values including following parameters:ANC:≥1.5x109/L, Platelet count:≥90x109/L, Hemoglobin:≥9.0 g/dL, Total bilirubin:≤1xULN, ALT and AST: ≤1.5xULN (for patients with liver metastases,ALT and AST:≤5xULN), ALP:≤2.5xULN, BUN and creatine:≤1xULN, creatine clearance rate:≥50 mL/min, LVEF:≥50%, QTcF:<450 ms (male), <470 ms (female),INR:≤1.5xULN, APTT:≤1.5xULN.
* Signed informed consent.

For subjects treated by Pyrotinib only:

- Failed or intolerable of prior therapies.

For subjects treated by Pyrotinib with Docetaxel:

- Failed or intolerable of prior therapies, no previous treatment of taxane, no previous treatment of HER2 targeted inhibitors.

Exclusion Criteria:

* Subjects with third space fluid that can not be controled by drainage or other methods.
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption.
* Steroid treatment for more than 50 days, or in need of long-term use of steroids.
* Less than 4 weeks from the last radiotherapy,chemotherapy，surgery，hermone treatment,target therapy, or less than 6 weeks from the nitrosoureas or mitomycin chemotherapy.
* Less than 4 weeks from the last clinical trial or adverse events of previous trials (not including alopecia or asthenia).
* Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
* Subjects who can not interrupt using of the drugs causing QT prolongation during study.
* Subjects with intracranial lesions (by MRI or CT).
* Subjects suffered from other malignancies during last 5 years, not including cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma.
* Subjects with bone or skin as the only target lesion.
* Receiving any other antitumor therapy.
* Known history of hypersensitivity to any of the components or metabolites of the investigational drugs or to Tween-80.
* Subjects with clear tendency of gastointestinal bleeding. Including the following: subjects with local active ulcer lesions and fecal occult blood (++) are excluded; subjects with less than 2 months from the last history of black stools or haematemesis are excluded; for subjects with fecal occult blood (+) and primary lesion not resected, endoscopy is required,if gastric ulcer is found and the principal investigator of the site consider possible occurence of gastointestinal bleeding, the subject should be excluded.
* Ongoing infection or peripheral neuropathy (determined by investigator).
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test or reluctant to take effective contraceptive measures throughout the trial period.
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study. Examples include, but are not limited to,hypertension, severe diabetes, or thyroid disease.
* Alcoholism, smoking (daily ≥ 5 roots) and other bad habits.
* Known history of neurological or psychiatric disease, including epilepsy or dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) of Pyrotinib and that of Pyrotinib with Docetaxel in patients with HER2 positive advanced gastric cancer | 21 days
  MTD will be defined as the maximum dose level at which no more than one subject out of three experience has a dose-limiting toxicity (DLT) upon completing one treatment cycle. DLT was defined as the certain AEs which were observed during the first cycle (D1-D21) of treatment

SECONDARY OUTCOMES:
Cmax of Pyrotinib and Pytotinib with Docetaxel in patients with HER2 positive advanced gastric cancer | 12 months
Tmax of Pyrotinib and Pytotinib with Docetaxel in patients with HER2 positive advanced gastric cancer | 12 months
T1/2 of Pyrotinib and Pytotinib with Docetaxel in patients with HER2 positive advanced gastric cancer | 12 months
AUCss of Pyrotinib and Pytotinib with Docetaxel in patients with HER2 positive advanced gastric cancer | 12 months
R of Pyrotinib and Pytotinib with Docetaxel in patients with HER2 positive advanced gastric cancer | 12 months
the number of participants with adverse event | 12 months
preliminary antitumor activity for the regimen | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Peking University, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Cancer center, Sun Yet-sen University, Guangzhou, Guangdong

REFERENCES:
- [Derived] Liu D, Kou F, Gong J, Wang Z, Zhang X, Li J, Li Y, Li J, Zhou J, Lu M, Wang X, Lu Z, Cao Y, Zou J, Zhu X, Xu R, Shen L. Pyrotinib alone or in combination with docetaxel in refractory HER2-positive gastric cancer: A dose-escalation phase I study. Cancer Med. 2023 May;12(9):10704-10714. doi: 10.1002/cam4.5830. Epub 2023 Apr 20. PMID 37081722
- [Derived] Chen Z, Xu Y, Gong J, Kou F, Zhang M, Tian T, Zhang X, Zhang C, Li J, Li Z, Lai Y, Zou J, Zhu X, Gao J, Shen L. Pyrotinib combined with CDK4/6 inhibitor in HER2-positive metastatic gastric cancer: A promising strategy from AVATAR mouse to patients. Clin Transl Med. 2020 Aug;10(4):e148. doi: 10.1002/ctm2.148. PMID 32898333